CLINICAL TRIAL: NCT04857762
Title: Anatomical Assessment Versus Pull Back REsting Full-cycle rAtio (RFR) Measurement for Evaluation of Focal and Diffuse Coronary Disease
Brief Title: Anatomical Assessment Versus Pull Back RFR Measurement
Acronym: READY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Szabolcs - Szatmár - Bereg County Hospitals and University Teaching Hospital, András Jósa Teaching H (Other)
Collaborators: Premier G Med Cardio Ltd. (Unknown)
Responsible Party: Principal Investigator, Zsolt Kőszegi, head of department, Szabolcs - Szatmár - Bereg County Hospitals and University Teaching Hospital, András Jósa Teaching H
Other Study IDs: 1292/2021
Record Dates: First submitted 2021-04-13; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Stenosis
Keywords: FFR, RFR
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The READY register is a multicenter open label registry of patients underwent invasive intracoronary FFR and RFR measurement using the Quantien system. The register collects clinical and epidemiological data of patients scheduled for invasive coronary physiology.

DETAILED DESCRIPTION:
Angiographic evaluation protocol:

Coronary diagnostic angiography is performed according to the routine clinical practice. The visual estimate of the diameters stenosis % of the culprit lesion(s) should be input prospectively in the modified Syntax segmentation scheme (https://coronart.hu/) where the corresponding ventricular segments supply is indicated on a polar map. On the same time, the operator is required to record characterize the coronary vessel disease as focal, diffuse or mixed type, and to document his plan for angioplasty on the basis of the visual assessment. The number and length of stents planned for implantation for each patient should be also documented on the basis of visual estimation before the physiological measurements.

Invasive coronary physiology assessment protocol:

PressurewireX will be advanced distally to the investigated lesion(s) of a coronary artery. Resting and hyperemic average pressures will be determined in this distal position (in FFR mode).

A resting manual pullback with 1-2 mm/s speed will be performed (in RFR mode) under simultaneous fluoroscopic control. The "store fluoro" option of the X-ray system allows the co-registration of the pressure drop(s) to the epicardial lesion(s) on the basis of the same time scale of the pullback and the stored fluoro. The use of marker(s) in the Quantien software can enhance the identification of the culprit interval(s) of the pressure pullback curve and the related angiographic details.

A substudy of the register is planned to achieve extended physiological assessment in patients with the suspicion of microvascular disease in line with the latest ESC guideline stressing the role of microcirculatory dysfunction in the adverse outcome events in patients with non-significant coronary stenoses by FFR (class IIa, level B recommendation).

According to the intracoronary average pressure values the pressure bounded CFR interval will be calculated (CFRpb). If the cut-off value CFR=2 lies inside the defined CFRpb interval, then a novel CFR calculation based on three-dimensional reconstruction and simple flow dynamic modelling will be performed to get the exact CFRp-3D value in order to diagnose or exclude microvascular disease. One simple possibility for the characterization of the microvasculature is to define the CFR/FFR index. This value below 2 indicate impaired microvascular vasodilator capacity. For getting more precise microvascular parameter, the flow modeling using the data of the 3D coronary reconstruction and the intracoronary pressure values will provide the microvascular resistance reserve (MRR).

Offline 3D angiographic reconstruction will be performed from the selected two angiograms of good quality, with at least 25◦ difference in angle, using dedicated 3D software.

Statistical Analysis:

Normal distribution will be tested. Descriptive statistics are planned as mean and SD, median (interquartile range), or counts (%) as appropriate. Categorical variables will be compared with the Pearson χ2test. Correlation among variables will be determined by calculating Spearman ρ correlation coefficient. All analyses will be performed in Medcalc program.

ELIGIBILITY:
Inclusion Criteria:

* At least one lesion on coronary artery branch greater than 2 mm in diameter assessed as 40-90% narrowing by visual estimation
* Invasive intracoronary FFR and RFR measurement using the Quantien system according to clinical decision

Exclusion Criteria:

* Patients with acute coronary syndrome
* Left main disease
* Contraindication for adenosine
* Coronary artery bypass graft on the investigated vessel
* Severe renal insufficiency (estimated glomerular filtration rate <30 ml/min/1.73 m2)
* Coronary angiography and pressure recordings not suitable for evaluation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease between 18-85 years.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Concordance of visual estimation and functional assessment | Baseline, before invasive functional assessment (The visual assessment is performed after the completion of the diagnostic coronary angiography, while the functional evaluation is recorded after the intracoronary physiological measurements)
  Comparison of the visual estimate of coronary lesions and the functional severity of the stenosis assessed by RFR pullback both on lesion- and vessel levels.
Characterization the coronary vessel for predominantly focal/diffuse or mixed type of the disease according to visual versus RFR pullback determination. | Baseline, before invasive functional assessment (The visual assessment is performed after the completion of the diagnostic coronary angiography, while the functional evaluation is recorded after the intracoronary physiological measurements)
  Focal disease: ∆RFR >0.05 for <25mm segment length (>0.002/mm) Diffuse disease: ∆RFR >0.05 for >25mm segment length If both focal and diffuse criteria are fulfilled in the investigated vessel, then mixed type disease is diagnosed
Evaluation of the concordance of the therapeutic strategies (conservative/PCI/CABG) on the basis of visual evaluation versus RFR measurements. | Baseline, pre-intervention (Theoretical clinical decision is made after the visual assessment of the diagnostic coronary angiography, while the final decision is made after the functional evaluation by intracoronary physiological measurements)
  Comparison of the rate of indication for the individual therapeutic strategies (conservative/PCI/CABG) by visual estimation and RFR measurements.

SECONDARY OUTCOMES:
In cases when the operator decides stent implantation, the planned number of stents also to be investigated according to the visual estimation versus RFR measurement. | Baseline, pre-intervention (Theoretical clinical decision is made after the visual assessment of the diagnostic coronary angiography, while the final decision is made after the functional evaluation by intracoronary physiological measurements)
  Comparison of the planned number of stents on the basis of visual estimation versus RFR measurement
In cases when the operator decides stent implantation, the total length of the planned stent(s) also to be investigated according to the visual estimation versus RFR measurement. | Baseline, pre-intervention (Theoretical clinical decision is made after the visual assessment of the diagnostic coronary angiography, while the final decision is made after the functional evaluation by intracoronary physiological measurements)
  Comparison of the length of the planned stent(s) on the basis of visual estimation versus RFR

CONTACTS AND LOCATIONS:
Locations (6):
- University Heart Center Graz, Division of Cardiology, Medical University Graz, Graz, Austria
- Hungary (5):
  - Department of Cardiology, Faculty of Medicine, University of Debrecen, Debrecen
  - Bacs-Kiskun County Hospital Recruiting Kecskemet, Hungary,, Kecskemét
  - Szabolcs - Szatmár - Bereg County Hospitals and University Teaching Hospital, András Jósa Teaching Hospital, Nyíregyháza
  - Heart Institute, Medical School, University of Pécs, Pécs
  - Invasive Cardiology Unit, Cardiology Center, University of Szeged, Szeged

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gould KL, Lipscomb K, Hamilton GW. Physiologic basis for assessing critical coronary stenosis. Instantaneous flow response and regional distribution during coronary hyperemia as measures of coronary flow reserve. Am J Cardiol. 1974 Jan;33(1):87-94. doi: 10.1016/0002-9149(74)90743-7. No abstract available. PMID 4808557
- [Background] Gould KL. Does coronary flow trump coronary anatomy? JACC Cardiovasc Imaging. 2009 Aug;2(8):1009-23. doi: 10.1016/j.jcmg.2009.06.004. PMID 19679290
- [Background] Beauman GJ, Vogel RA. Accuracy of individual and panel visual interpretations of coronary arteriograms: implications for clinical decisions. J Am Coll Cardiol. 1990 Jul;16(1):108-13. doi: 10.1016/0735-1097(90)90465-2. PMID 2358583
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Patel MR, Calhoon JH, Dehmer GJ, Grantham JA, Maddox TM, Maron DJ, Smith PK. Correction to: ACC/AATS/AHA/ASE/ASNC/SCAI/SCCT/STS 2017 Appropriate Use Criteria for Coronary Revascularization in Patients With Stable Ischemic Heart Disease. J Nucl Cardiol. 2018 Dec;25(6):2191-2192. doi: 10.1007/s12350-018-1292-x. PMID 29748874
- [Background] Jeremias A, Davies JE, Maehara A, Matsumura M, Schneider J, Tang K, Talwar S, Marques K, Shammas NW, Gruberg L, Seto A, Samady H, Sharp A, Ali ZA, Mintz G, Patel M, Stone GW. Blinded Physiological Assessment of Residual Ischemia After Successful Angiographic Percutaneous Coronary Intervention: The DEFINE PCI Study. JACC Cardiovasc Interv. 2019 Oct 28;12(20):1991-2001. doi: 10.1016/j.jcin.2019.05.054. PMID 31648761
- [Background] Warisawa T, Cook CM, Howard JP, Ahmad Y, Doi S, Nakayama M, Goto S, Yakuta Y, Karube K, Shun-Shin MJ, Petraco R, Sen S, Nijjer S, Al Lamee R, Ishibashi Y, Matsuda H, Escaned J, di Mario C, Francis DP, Akashi YJ, Davies JE. Physiological Pattern of Disease Assessed by Pressure-Wire Pullback Has an Influence on Fractional Flow Reserve/Instantaneous Wave-Free Ratio Discordance. Circ Cardiovasc Interv. 2019 May;12(5):e007494. doi: 10.1161/CIRCINTERVENTIONS.118.007494. PMID 31084237
- [Background] Svanerud J, Ahn JM, Jeremias A, van 't Veer M, Gore A, Maehara A, Crowley A, Pijls NHJ, De Bruyne B, Johnson NP, Hennigan B, Watkins S, Berry C, Oldroyd KG, Park SJ, Ali ZA. Validation of a novel non-hyperaemic index of coronary artery stenosis severity: the Resting Full-cycle Ratio (VALIDATE RFR) study. EuroIntervention. 2018 Sep 20;14(7):806-814. doi: 10.4244/EIJ-D-18-00342. PMID 29790478
- [Background] Van't Veer M, Pijls NHJ, Hennigan B, Watkins S, Ali ZA, De Bruyne B, Zimmermann FM, van Nunen LX, Barbato E, Berry C, Oldroyd KG. Comparison of Different Diastolic Resting Indexes to iFR: Are They All Equal? J Am Coll Cardiol. 2017 Dec 26;70(25):3088-3096. doi: 10.1016/j.jacc.2017.10.066. PMID 29268922
- [Background] Hoshino M, Yonetsu T, Sugiyama T, Kanaji Y, Hamaya R, Kanno Y, Hada M, Yamaguchi M, Sumino Y, Usui E, Hirano H, Horie T, Nogami K, Ueno H, Misawa T, Murai T, Lee T, Kakuta T. All Resting Physiological Indices May Not Be Equivalent - Comparison Between the Diastolic Pressure Ratio and Resting Full-Cycle Ratio. Circ J. 2020 Jun 25;84(7):1147-1154. doi: 10.1253/circj.CJ-19-1110. Epub 2020 Jun 4. PMID 32493861
- [Derived] Koszegi Z, Berta B, Toth GG, Tar B, Uveges A, Agoston A, Szucs A, Szabo GT, Barta J, Szuk T, Czuriga D, Komocsi A, Ruzsa Z. Anatomical Assessment vs. Pullback REsting full-cycle rAtio (RFR) Measurement for Evaluation of Focal and Diffuse CoronarY Disease: Rationale and Design of the "READY Register". Front Cardiovasc Med. 2021 Dec 13;8:784220. doi: 10.3389/fcvm.2021.784220. eCollection 2021. PMID 34966799